CLINICAL TRIAL: NCT06404775
Title: External Mastalgia-oil Versus Oral Tamoxifen in Premenopausal Women with Severe Mastalgia: a Double-blind, Double-simulated, Positive-controlled Randomized Clinical Trial
Brief Title: External Mastalgia-oil Versus Oral Tamoxifen in Premenopausal Women with Severe Mastalgia
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Chang Gong, Clinical Professor, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYSKY-2024-292-02
Record Dates: First submitted 2024-04-26; First posted 2024-05-08 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Mastalgia
MeSH Terms: conditions — Mastodynia | interventions — Tamoxifen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- external mastalgia-oil plus oral tamoxifen placebo (Experimental)
  Interventions: Drug: mastalgia-oil, tamoxifen placebo
- oral tamoxifen plus external mastalgia-oil placebo (Active Comparator)
  Interventions: Drug: mastalgia-oil placebo, tamoxifen

INTERVENTIONS:
Drug: mastalgia-oil, tamoxifen placebo — external mastalgia-oil 1 ml/d per breast plus oral tamoxifen placebo 10mg/d for 3 consecutive menstrual cycles
  Arms: external mastalgia-oil plus oral tamoxifen placebo
Drug: mastalgia-oil placebo, tamoxifen — oral tamoxifen 10mg/d plus external mastalgia-oil placebo 1 ml/d per breast for 3 consecutive menstrual cycles
  Arms: oral tamoxifen plus external mastalgia-oil placebo

SUMMARY:
This is a single-center, double-blind, double-simulated, positive-controlled, randomized clinical trial to explore the efficacy and safety of external mastalgia-oil versus oral tamoxifen in premenopausal women with severe mastalgia.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal females aged ≥ 18 years old
* Pre-existing regular menstrual cycle (28 ± 3 days) with mastalgia lasting for at least 6 consecutive menstrual cycles; with severe mastalgia [visual analog scale (VAS) score ≥ 4 for at least 7 days] and without chest wall pain in the baseline menstrual cycle (nonmedicated menstrual cycle)
* With breast ultrasound: BI-RADS classification 1-3; if mammography is required: also BI-RADS classification 1-3
* Willingness to follow up and complete required tests; ability to complete questionnaires independently or with assistance
* Willingness to use effective contraception (vaginally administered estrogen and hormone-coated IUDs are permitted) prior to study entry, during study participation, and for three months after discontinuation of the drug; negative pregnancy test in females of childbearing potential
* Requisite laboratory values:white blood cell count: ≥ 4.0 × 10^9/L, absolute neutrophil count: ≥ 2 × 10^9/L, platelet count: ≥ 100 × 10^9/L; hemoglobin: ≥ 110 g/L; aspartate aminotransferase and alanine aminotransferase: ≤ upper limit of normal, alkaline phosphatase: ≤ upper limit of normal, blood total bilirubin: ≤ upper limit of normal; serum creatinine and blood urea nitrogen: ≤ upper limit of normal

Exclusion Criteria:

* With suspected breast disease (e.g., mastitis, malignant breast tumor) other than breast pain or benign breast cysts, or with other malignant tumors
* Use of hormonal medications (e.g., oral contraceptives, glucocorticoids, etc.), sex hormone modulators (SERMS, AIs, SERDs, etc.), B vitamins, essential oils, nonsteroidal anti-inflammatory drugs, or higher pain relievers in the past 3 months; use of tamoxifen or analogs in the past 6 months
* Prior history of breast surgery (including minimally invasive surgery), history of malignancy, or history of thromboembolism within the last 5 years (history of varicose veins and superficial phlebitis allowed)
* Smokers; tamoxifen or essential oils systemic/skin sensitization
* With serious primary diseases of the heart, liver, kidneys and hematopoietic system, or mental illness, etc.
* Accompanied by skin damage on the breast that destroys the stratum corneum (e.g., eczema, ulcers)
* Serious or uncontrolled infections that may interfere with study treatment or assessment of study results, including but not limited to active hepatitis viral infection, human immunodeficiency virus antibody positivity, syphilis spirochete antibody positivity with evidence of active infection, and pulmonary infections
* Subjects who are breastfeeding or pregnant at the time of screening (of childbearing age and with serum human chorionic gonadotropin test results higher than the reference value); subjects of childbearing age who have had unprotected sex with a heterosexual partner within 2 weeks prior to the screening; subjects of childbearing age who are planning to prepare for conception, become pregnant, breastfeed, or donate their eggs during the test period or within 3 months of the end of the test; and those with implanted breasts
* Decrease in total breast pain score by more than 25% during the placebo lead-in cycle. These patients will not receive subsequent randomization and treatment.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 456 (Estimated)
Dates: Start 2025-01-16 (Estimated); Primary Completion 2029-01-16 (Estimated); Study Completion 2030-05-16 (Estimated)

PRIMARY OUTCOMES:
Mastalgia clinical response rate | Within 4 weeks after the end of the third treatment menstrual cycle
  The recruited patients with mastalgia will be asked to record their symptoms of breast pain using a daily VAS breast pain chart, and the sum of the daily VAS within a menstrual cycle is considered the breast pain score (BPS). Effective rate (%)= [BPS (P) - BPS (T3)]/BPS (P)*100%, where BPS (P) indicates BPS of the placebo lead-in cycle and BPS (T3) indicates BPS at the end of the third treatment cycle. An effective rate of more than 50% is considered a clinical response.
Safety (adverse events) | from signing the informed consent form until 4 weeks after the end of the third treatment menstrual cycle
  Total incidence of the following adverse events: hot flashes + leukorrhea + menorrhagia + nausea + headache + skin reactions. Adverse events will be assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events (version 5.0).Each patient will be counted only once for the above adverse events experienced.

SECONDARY OUTCOMES:
Subgroup mastalgia clinical response rate | Within 4 weeks after the end of the third treatment menstrual cycle
  Mastalgia clinical response rate in women with cyclical mastalgia; Mastalgia clinical response rate in women with non-cyclical mastalgia
Breast nodularity | Within 7 days before the first treatment and the end of each treatment menstrual cycle
  Breast nodularity will be assessed according to the Lucknow-Cardiff breast nodularity scale.The above breast nodularity scale is a 5-point ordinal scale depicting increasing order of nodularity in upper outer quadrants of the breasts. Grade-0 depicts a smooth textured breast with extreme extent of normalcy and grade-4 the maximum nodularity.
Pharmacokinetics of mastodynia-oil | Within 4 weeks after the end of the third treatment menstrual cycle
  Collection of blood samples for pharmacokinetic trough concentration-effect analysis of mastodynia-oil
Changes in blood biochemical indicators | Within 4 weeks after the end of the third treatment menstrual cycle
  Tamoxifen-specific indicators: estradiol, progesterone, et al. and their correlation with the primary endpoints were detected in blood before and after treatment using ELISA.
Changes in blood metabolites | Within 4 weeks after the end of the third treatment menstrual cycle
  Comparison of changes in blood metabolites before and after treatment and their correlation with primary endpoints using metabolomics.

CONTACTS AND LOCATIONS:
Overall Officials: Chang Gong, Prof, Principal Investigator — Breast Tumor Center, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kumar S, Rai R, Das V, Kumar S, Dwivedi V, Agrawal GG. Visual analogue scale for assessing breast nodularity in non-discrete lumpy breasts: the Lucknow-Cardiff breast nodularity scale. Breast. 2010 Jun;19(3):238-42. doi: 10.1016/j.breast.2010.02.002. Epub 2010 Mar 11. PMID 20223665